CLINICAL TRIAL: NCT01496326
Title: A Pilot Study to Compare the Efficacy and Safety of a Novel 10% Ibuprofen Formulation Versus Placebo Alone Applied to the Knee in Patients With Painful Osteoarthritis of the Knee
Brief Title: Osteoarthritis Topical Treatment
Acronym: ANTIPAIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioChemics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BC-IBU-CH-001
Record Dates: First submitted 2011-12-15; First posted 2011-12-21 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; knee pain
MeSH Terms: conditions — Osteoarthritis | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ibuprofen (Experimental)
  Interventions: Drug: Ibuprofen
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ibuprofen — 10% ibuprofen cream formulation at a dose of 200mg
  Arms: Ibuprofen
Drug: placebo — 2 grams of placebo cream for 14 days
  Arms: Placebo

SUMMARY:
This is a phase 2a clinical trial performed to evaluate the efficacy of a topical treatment of ibuprofen compared to the use of a placebo topical treatment.

A multi-center, double-blinded, randomized placebo controlled study. Study length: 14 days Dosing twice daily (b.i.d.)

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female patients aged at least 40 years.
* Primary osteoarthritis in a single knee joint, grade II/III based on the Kellgren and Lawrence classification system.
* Radiographic evidence consistent with osteoarthritis carried out within 6 months before screening.
* pain is currently not adequately controlled with a simple analgesic or an NSAID OR would necessitate treatment, but is not yet treated.

Main Exclusion Criteria:

* Concomitant presence of another type of continuous pain that is more severe in intensity in comparison with the osteoarthritis target joint pain
* Osteoarthritis causing significant pain in any joint other than the identified knee, or contralateral knee (≥ 20 mm pain) as confirmed by a separate VAS at visit 1 for any other painful joint concerned.
* Female patients who are pregnant or breast-feeding.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) Pain scale | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Carter, Ph.D., Study Director — BioChemics, Inc.
Locations (4):
- Switzerland (4):
  - Sankt Gallen
  - Schaffhausen
  - Zurich
  - Rheumaklinik und Institut für Physikalische Medizin Universitätsspital, Zurich

REFERENCES:
- [Derived] Varadi G, Zhu Z, Blattler T, Hosle M, Loher A, Pokorny R, Frey D, Carter SG. Randomized clinical trial evaluating transdermal Ibuprofen for moderate to severe knee osteoarthritis. Pain Physician. 2013 Nov-Dec;16(6):E749-62. PMID 24284856